CLINICAL TRIAL: NCT03683043
Title: Comparative Study Between ICSI Results in Transvaginal Ultrasound Guided Embryo Transfer and Transabdominal Ultrasound Guided Embryo Transfer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 40
Record Dates: First submitted 2018-09-19; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Invitro Fertilization
MeSH Terms: interventions — Leuprolide; Embryo Transfer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transabdominal guided transfer (Active Comparator): In the trans-abdominal guided embryo transfer group, the patients' bladder were filled by 500-700 ml saline; in order to enhance the visualization. The trans-abdominal probe is applied on pelvis by an assistant nurse or the attending gynecologist intern
  Interventions: Drug: Long GnRH agonist protocol; Procedure: Embryo transfer
- Transvaginal guided transfer (Active Comparator): the trans-vaginal guided embryo transfer group had their bladder emptied by the gynecologist via catheter prior to transfer or else the patient was asked to void. The speculum is applied followed by insertion of the outer sheath of the transfer catheter. The speculum is removed with caution; to maintain the outer sheath in place. The TVUS probe is applied vaginally and endometrium is visualized before transfer. The transfer is done through an inner catheter applied to the already inserted outer sheath
  Interventions: Drug: Long GnRH agonist protocol; Procedure: Embryo transfer

INTERVENTIONS:
Drug: Long GnRH agonist protocol — 8. The patients follow long protocol, which includes down regulation starting on day 21 of the previous cycle. The patient is seen after 14 days to confirm down regulation. Serum E2 ≤ 50 pg/ mL and no ovarian cysts observed in transvaginal US.
  9. Induction is started on day 3 of the current cycle by gonadotrophins (FSH and LH) daily IM or SC injections provided that the different preparations at the market can be used.
  Other Names: Leuprolide acetate ( Lupron)
Procedure: Embryo transfer — Cusco speculum was used to allow access to the cervix. The vagina was flushed by saline, and the cervical mucus is removed by Q-tips and/ or suction tubes. In few cases, where patients had long vaginae; two Sims' speculums were used to spread the vaginal anterior and posterior vaginal walls apart. In these cases, the attending nurse assisted the gynecologists during transfer The gynecologist asks the embryologist to load the embryos in the transfer catheter, and the gynecologist receives the loaded catheter from a window connecting the lab and operating room. In cases of trans-vaginal ultrasound guided embryo transfer the embryologist hands in the catheter to the gynecologists in the outer sheath and the gynecologist injects slowly the fluid containing the embryo/s. All patients are asked to rest for 30 minutes after the transfer

SUMMARY:
This prospective study will be conducted on 120 patients candidates for ICSI cycle and following the long protocol for controlled ovarian stimulation; the patients were randomly allocated in a 1:1 ratio to either group A; where the embryo transfer was assisted by transabdominal ultrasound and group B; where the embryo transfer was assisted by Transvaginal ultrasound. The study nurse opened the sealed envelopes according to sequence of attendance of patients to allocate patients to the assigned group. Both the patient and the operator were blind to the assigned group.

All the transfers were done on day 3 after OPU for at least 2 grade I embryos using the Edwards-Wallace embryo replacement catheter using the same ultrasound device. Quantitative serum hCG test was done for all patients 14 days after the transfer.

DETAILED DESCRIPTION:
One hundred and twenty patients were randomly allocated to either the trans-abdominal guided embryo transfer group (n= 60) or the transvaginal guided embryo tranfer group ( n = 60) . The investigators used a computer generated randomization table obtained from http://graphpad. com/quickcalcs/randomize1 and sequentially numbered sealed opaque envelopes to randomize the patients to the study groups. The allocation information was written on a card placed in the sealed envelopes. A colleague (who was not directly involved in the study) prepared the randomization table and the sealed envelopes.The patients were blind to the assigned group. The gynecologists were as well blind to the received treatment.

Patients included in the study are consenting to controlled ovarian hyperstimulation protocol, folliculometery visits, ovarian stimulation medications, ovum pick up, embryo transfer, luteal phase support, possible complications, as well as consenting to disclosure of pregnancy test results 14 days after embryo transfer.

After obtaining an informed written consent, each patient will be submitted to the following:

1. Full history taking including: name, age, menstrual history, history of previous trials (if any), obstetric history, medical history, and labs.
2. The husband's history and andrologist consultation -if any- are revised. All cases of severe male factor were excluded.
3. Clinical examination including: vital signs, weight, height, abdominal examination are done and recorded in the patient's sheet.
4. TVUS to assess the uterus, adnexa, cul-de-sac for any abnormalities and the antral follicular count is assessed on day 2-5 of the cycle and recorded.
5. All patients do serum FHS, LH, E2, Prolactin, TSH on D2 or D3 of the menstrual cycle.
6. Fasting and 2 hours post prandial blood sugar, HBsAg, and HCV antibodies, liver and kidney functions test are done for all patients prior to ovum pick up and to be revised by both the gynecologist and the anesthesiologist.
7. All the previous data are recorded in the patient's sheet at first visit. Folliculometery is done and recorded - in addition to any new findings- every visit. Uterine congenital anomalies and uterine pathologies seen by ultrasound are recorded.
8. The patients follow long protocol, which includes down regulation starting on day 21 of the previous cycle. The patient is seen after 14 days to confirm down regulation. Serum E2 ≤ 50 pg/ mL and no ovarian cysts observed in transvaginal US.
9. Induction is started on day 3 of the current cycle by gonadotrophins (FSH and LH) daily IM or SC injections provided that the different preparations at the market can be used. The number of ampoules given per dose is determined by infertility consultant.
10. The duration of induction ranges from 10-14 days, during which the patient is assessed by TVUS in each folliculometery visit; to assess the rate of growth and the endometrium.
11. When the majority of cohort of follicles reach 18-22 mm, hCG trigger 5000-10000 IU is administered IM and the ovum pick up is done 34-36 hours later.
12. The OPU procedure is done at the operation room under total aseptic conditions, and the patient receives sedation by anethiologist prior to the procedure.
13. OPU is done while the patient is in lithotomy position by inserting the TVUS probe with the needle guide attached to it in the lateral fornices of the vagina. The needle is connected to a suction device; which operates to create negative pressure for collection of the follicular fluid in tubes.
14. The tubes are handed in to the nurse and in turn the nurse hands it in to the embryologist via a window in the operation room connected to the embryology lab.
15. M2 cells of the collected ova are cultured and injected by sperms under electron microscope. Division takes place in the following 24 hours and only 'Grade 1' and 'Grade 2' embryos are transferred on D3.
16. The patient receives luteal phase support; progesterone 400 mg suppositories twice daily starting from the day of OPU.
17. Embryos are commonly transferred on day 3 after OPU. The endometrium thickness and echogenicity are checked prior to ET.
18. All the embryos transferred on day of ET are re assessed by the embryologist to determine their grade.
19. Embryos were scored for three parameters on day 2 (41-44 h after insemination/injection) and again on day 3 (66-71 h post-insemination/injection): (i) fragmentation (GI = no fragmentation, GII = 20% or less by volume of anucleated fragments); (ii) number of blastomeres; (iii) number of multinucleated blastomeres.
20. In both groups, Cusco speculum was used to allow access to the cervix. The vagina was flushed by saline, and the cervical mucus is removed by Q-tips and/ or suction tubes. In few cases, where patients had long vaginae; two Sims' speculums were used to spread the vaginal anterior and posterior vaginal walls apart. In these cases, the attending nurse assisted the gynecologists during transfer.
21. In the trans-abdominal guided embryo transfer group, the patients' bladder were filled by 500-700 ml saline; in order to enhance the visualization. The trans-abdominal probe is applied on pelvis by an assistant nurse or the attending gynecologist intern.
22. While the trans-vaginal guided embryo transfer group had their bladder emptied by the gynecologist via catheter prior to transfer or else the patient was asked to void. The speculum is applied followed by insertion of the outer sheath of the transfer catheter. The speculum is removed with caution; to maintain the outer sheath in place. The TVUS probe is applied vaginally and endometrium is visualized before transfer. The transfer is done through an inner catheter applied to the already inserted outer sheath.
23. In all patients of the two groups the Edwards-Wallace embryo replacement catheter was used. And ultrasound device used during folliculometery, OPU, and ET was Mindray DP-5/ Shenzen- China. The probe frequency 2.0/3.5/5.0/6.0/H4.6/H6.0MHz
24. The gynecologist asks the embryologist to load the embryos in the transfer catheter, and the gynecologist receives the loaded catheter from a window connecting the lab and operating room. In cases of trans-vaginal ultrasound guided embryo transfer the embryologist hands in the catheter to the gynecologists in the outer sheath and the gynecologist injects slowly the fluid containing the embryo/s.
25. All patients are asked to rest for 30 minutes after the transfer
26. The intensity of pain was measured using a visual analog scale (VAS). Visual analog scale was a horizontal line, 100 mm in length, anchored by word descriptors at each end (0 = the absence of pain; 100 = the worst experienced pain). The patients were asked to mark on the line the point that represented their perception of pain. The VAS score was determined by measuring in millimeters from the left hand end of the line to the point that the patient marked. The patients were asked to evaluate the intensity of pain during and 30 minutes after the procedure (Fouda et al, 2016)
27. At the end of the procedure the operator was asked to comment on the over all technique of embryo transfer by TAUS or TVUS, whether easy or difficult regardless the difficulty or ease of passage of transfer catheter through the cervix.
28. The operator also recorded the quality of visualization in the transfer sheet whether good or fair.
29. All patients are prescribed to the same luteal phase support regimen by progesterone 400 mg vaginal suppositories twice daily.
30. Quantitative serum hCG is measured 14 days after ET for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Infertile female patients aged 20-37 years old undergoing IVF
* Long protocol
* Embryo transfer of fresh cycles D3

Exclusion Criteria:

* Uterine abnormalities e.g. sub-mucous fibroid, or fibroids indenting the endometrium, polyps, Ashermann, etc.
* Poor responders
* Female patients ˃35 years old
* Medical disorders e.g. DM, HTN
* Immunological disorders e.g. SLE, APS
* Cervical distortions
* Thyroid or adrenal dysfunction
* Endometriosis grade 3 or 4

Ages: 19 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 14 days after embryo transfer
  detection of intrauterine gestational sac using transvaginal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed maged, MD, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided